CLINICAL TRIAL: NCT06158919
Title: A Phase II Clinical Study of PD-1 Inhibitors Combined With Fruquintinib and Chemotherapy in First-line Treatment of HER2-negative Advanced G/GEJ Cancer
Brief Title: A Study of PD-1 Inhibitors Combined With Fruquintinib and Chemotherapy in First-line Treatment of HER2-negative Advanced G/GEJ Cancer
Acronym: G/GEJ cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, Medical oncology chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-FIX
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer/Adenocarcinoma of Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 Inhibitors Combined With Fruquintinib and Chemotherapy (Experimental): Combined treatment period: A total of 6 cycles of combined treatment Fruquintinib: 4 mg/d, qd po, d1-14, q3w. Nivolumab: 360mg iv.gtt d1, q3w or Sindilizumab: 200mg iv.gtt d1, q3w SOX: Oxaliplatin 130mg/m2 iv.gtt d1, Teysuno 40mg/m2 p.o.b.i.d. d1~ 14q3w. Or XELOX regimen: oxaliplatin 130mg/m2 iv.gtt d1 Capecitabine 1000mg/m2 p.o. b.i.d. d1~ 14q3w.
  Maintenance treatment period:
  Fruquintinib: 4 mg/d, qd po, d1-14, q3w. Nivolumab: 360mg iv.gtt d1, q3w or Sindilizumab: 200mg iv.gtt d1, q3w Teysuno 40mg/m2 p.o.b.i.d. d1~14 q3w or Capecitabine 1000mg/m2 p.o.b.i.d. d1~14 q3w.
  Maintenance of treatment until disease progression or toxicity becomes intolerable.The longest duration of PD-1 inhibitor treatment is 24 months.
  Interventions: Drug: Fruquintinib、Nivolumab、Sintilimab、Oxaliplatin、Teysuno、Capecitabine

INTERVENTIONS:
Drug: Fruquintinib、Nivolumab、Sintilimab、Oxaliplatin、Teysuno、Capecitabine — Combined treatment period: A total of 6 cycles of combined treatment Fruquintinib: 4 mg/d, qd po, d1-14, q3w. Nivolumab: 360mg iv.gtt d1, q3w or Sintilimab: 200mg iv.gtt d1, q3w SOX : Oxaliplatin 130mg/m2 iv.gtt d1, Teysuno 40mg/m2 p.o.b.i.d. d1~ 14q3w. Or XELOX regimen: oxaliplatin 130mg/m2 iv.gtt d1 Capecitabine 1000mg/m2 p.o. b.i.d. d1~ 14q3w.
  Maintenance treatment period:
  Fruquintinib: 4 mg/d, qd po, d1-14, q3w. Nivolumab: 360mg iv.gtt d1, q3w or Sintilimab: 200mg iv.gtt d1, q3w Teysuno 40mg/m2 p.o.b.i.d. d1~14 q3w or Capecitabine 1000mg/m2 p.o.b.i.d. d1~14 q3w.
  Maintenance of treatment until disease progression or toxicity becomes intolerable.

SUMMARY:
This is an open-label, single-arm, single-center clinical study to investigate the safety and efficacy of fuquinitinib combined with PD-1 inhibitors and first-line chemotherapy in the treatment of inoperable HER2-negative advanced GC/GEJC.

Eligible enrolled patients received 6 cycles of combined treatment with fuquinitinib combined with PD-1 inhibitor and chemotherapy (XELOX/SOX) regimen. Maintenance treatment was fuquinitinib combined with PD-1 inhibitor and Teghio/capecitabine until disease progression or toxicity became intolerable. The longest duration of PD-1 inhibitor treatment is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;

2.18-80 years old (including 18 and 80 years old), male or female;

3. Patients with unresectable advanced or metastatic gastric/esophagogastric junction adenocarcinoma confirmed by pathology or histology;

4.ECOG physical status 0-1

5. Expected survival ≥3 months;

6. Have not received any anti-tumor therapy (including chemotherapy, targeted therapy, immunotherapy, etc.) for unresectable advanced or metastatic gastric cancer; If you have received adjuvant therapy after radical gastrectomy of gastric cancer, it is required that the time between the discovery of metastatic disease and the end of the last adjuvant chemotherapy is greater than 6 months);

7. Must have at least one measurable lesion (meet the RECIST v1.1 standard);

8. The functions of vital organs meet the following requirements (the use of any blood components and cell growth factors is not allowed within the first 14 days of enrollment) :

* Absolute neutrophil count ≥1.5×109/L, white blood cell ≥3.0×109/L;

  * Platelet ≥90×109/L;

    * Hemoglobin ≥8g/dL;

      * Total bilirubin TBIL≤1.5 times ULN;

        ⑤ALT and AST≤2.5 times ULN;

        ⑥ Urea/urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN (and creatinine clearance (CCr) ≥ 50mL/min);

        ⑦Left ventricular ejection fraction (LVEF) ≥50%;

        ⑧Fridericia Corrected QT Interval (QTcF) <470 milliseconds;

        ⑨INR≤1.5 x ULN, APTT≤1.5 x ULN;

        ⑩Thyroid function, thyroid stimulating hormone (TSH) ≤ upper limit of normal (ULN), if abnormal FT3 and FT4 levels should be examined, FT3 and FT4 levels can be included if normal;

        9. Premenopausal and postmenopausal women < Women of 1 year must have a negative serum or urine pregnancy test before treatment.

Exclusion Criteria:

* 1. Patients with known HER-2 status (immunohistochemical 3+, or immunohistochemical 2+&FISH positive);

  2. Had other malignancies within 5 years prior to admission, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;

  3. Previously received allogeneic bone marrow transplantation or organ transplantation;

  4. Severe cardiovascular disease, including unstable angina pectoris or myocardial infarction, in the 6 months prior to enrollment;

  5. Subjects who are allergic to the investigational drug or any of its adjuncts;

  6. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg;

  7. Had any disease or condition affecting drug absorption before enrollment, or the patient could not take drugs orally;

  8. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unexcised tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;

  9. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months >30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks >5 mL of fresh blood) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;

  10. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure >Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) <50%;

  11. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);

  12. Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (≥1×104 copies /mL or >2000 IU/ mL); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL);

  13. The patient has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; The patient had vitiligo; Those with complete remission of asthma in childhood can be included without any intervention in adulthood; Patients with asthma requiring medical intervention with bronchodilators are not included); Replacement therapy is not considered systemic, and the following patients may be included: have a history of autoimmune related hypothyroidism and are receiving thyroid hormone replacement therapy; Type 1 diabetes can be controlled by insulin therapy.

  14. Immunosuppressive use of immunosuppressants or systemic hormone therapy within 7 days prior to enrollment for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormone).

  15. Currently suffering from interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, radiation pneumonia;

  16. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;

  17. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;

  18. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume ≥1.0g;

Patients considered inappropriate for inclusion in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival

SECONDARY OUTCOMES:
ORR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Objective response rate
DCR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  disease control rate
OS | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhu, Principal Investigator — Fudan University
Locations (1):
- Fudan University ShangHai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No